CLINICAL TRIAL: NCT02453087
Title: An Open-label, Multicenter, Phase 1/1b Dose Escalation Study Evaluating the Pharmacokinetics, Safety, Tolerability, and Preliminary Efficacy of DCDS0780A, Alone or in Combination With Rituximab, or Obinutuzumab, in Patients With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Study of Escalating Doses of DCDS0780A in Participants With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29687
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DCDS0780A Monotherapy (Experimental): Participants will receive escalating doses of DCDS0780A as intravenous infusion as monotherapy on Day 1 of each 21-day cycle up to approximately 1 year or until disease progression or unacceptable toxicity (whichever comes first).
  Interventions: Drug: DCDS0780A
- DCDS0780A + Rituximab (Experimental): Participants will receive escalating doses of DCDS0780A on Day 2 of Cycles 1 and 2, and from Cycle 3 onwards on Day 1 of each 21-day cycle in combination with rituximab at a dose of 375 milligrams per square meter (mg/m^2) of body surface area as intravenous infusion on Day 1 of each 21-day cycle up to approximately 1 year or until disease progression or unacceptable toxicity (whichever comes first).
  Interventions: Drug: DCDS0780A; Drug: Rituximab
- DCDS0780A + Obinutuzumab (Experimental): Participants will receive escalating doses of DCDS0780A on Day 2 of Cycles 1 and 2, and from Cycle 3 onwards on Day 1 of each 21-day cycle in combination with obinutuzumab at a dose of 1000 milligrams (mg) as intravenous infusion on Days 1, 8, and 15 of Cycle 1, and from Cycle 2 onwards on Day 1 of each 21-day cycle up to approximately 1 year or until disease progression or unacceptable toxicity (whichever comes first).
  Interventions: Drug: DCDS0780A; Drug: Obinutuzumab

INTERVENTIONS:
Drug: DCDS0780A — Participants will receive escalating doses of DCDS0780A as intravenous infusion.
Drug: Rituximab — Participants will receive rituximab at a dose of 375 mg/m^2 of body surface area as intravenous infusion.
  Other Names: Rituxan®; MabThera®
  Arms: DCDS0780A + Rituximab
Drug: Obinutuzumab — Participants will receive obinutuzumab at a dose of 1000 milligrams (mg) as intravenous infusion.
  Other Names: GA101; Gazyva™; Gazyvaro™
  Arms: DCDS0780A + Obinutuzumab

SUMMARY:
This open-label, multicenter, Phase 1/1b study will evaluate the safety, tolerability, and pharmacokinetics of increasing doses of DCDS0780A in participants with relapsed or refractory B-cell non-Hodgkin's lymphoma. In the combination portion of the study, the safety and tolerability of DCDS0780A in combination with rituximab or obinutuzumab will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Histologically confirmed B-cell non-Hodgkin's lymphoma that has relapsed after or failed to respond to at least one prior treatment regimen and for which no suitable therapy of curative intent or higher priority exists
* A clinical indication for treatment as determined by the investigator
* Availability of archival or freshly collected tumor tissue before study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Fasting (greater than or equal to [>=] 8 hours) glucose less than or equal to (<=) 160 milligrams per deciliter (mg/dL)
* Participants requiring anti-diabetic medications must be on a stable dose and regimen for >=4 weeks
* Adequate hematologic function without growth factor or transfusion support
* For women who are not postmenopausal (>= 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods as specified in protocol
* For men: agreement to remain abstinent or use a condom plus an additional contraceptive method as specified in protocol

Exclusion Criteria:

* Prior use of any monoclonal antibody or antibody-drug conjugate within 4 weeks before Cycle 1, Day 1
* Treatment with radiotherapy, any chemotherapeutic agent, systemic steroids used as an anti-neoplastic agent, or any other investigational anti-cancer agent within 2 weeks prior to Cycle 1, Day 1
* Completion of autologous stem cell transplant within 100 days prior to Cycle 1, Day 1
* Prior allogeneic stem cell transplant
* Current or history of CNS lymphoma
* Current Grade greater than (>) 1 toxicity (except alopecia and anorexia) from prior therapy
* Current Grade >1 peripheral neuropathy from any cause
* Glycosylated hemoglobin (HbA1c) >=7.5 percent (%)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Prior irradiation to lung fields
* Clinically significant pulmonary disease
* Recent major surgery within 4 weeks prior to Cycle 1, Day 1, other than superficial lymph node biopsies for diagnosis
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Presence of positive test results for hepatitis B (hepatitis B surface antigen [HbsAg] and/or total hepatitis B core antibody [anti-HBc]) or hepatitis C (hepatitis C virus [HCV] antibody)
* Known history of human immunodeficiency virus (HIV) seropositive status
* Women who are pregnant or lactating or intending to become pregnant during the study
* Any abnormal laboratory values as specified in protocol
* Requirement for any excluded medication as specified in protocol
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications, including inadequately controlled diabetes or significant cardiovascular disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* Participants in Phase 1b Stage Only: Vaccination with live vaccines within 6 months before Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Baseline up to 30 days after the last dose of study drug (up to 1 year)
Percentage of Participants with Dose-Limiting Toxicities | Days 1 to 21
Maximum Tolerated Dose (MTD) of DCDS0780A | Days 1 to 21
Recommended Phase 2 Dose (RP2D) of DCDS0780A | Days 1 to 21

SECONDARY OUTCOMES:
Area Under the Serum Concentration-Time Curve (AUC) for DCDS0780A Total Antibody | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to end of treatment (ET) visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Maximum Observed Serum Concentration (Cmax) for DCDS0780A Total Antibody | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Total Clearance (CL) of DCDS0780A Total Antibody | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Half-life (t1/2) of DCDS0780A Total Antibody | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Volume of Distribution Under Steady-State Conditions (Vss) of DCDS0780A Total Antibody | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Area Under the Plasma Concentration-Time Curve (AUC) for DCDS0780A Conjugate (Antibody-Conjugated Monomethyl Auristatin E [acMMAE]) | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Maximum Observed Plasma Concentration (Cmax) for acMMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Total Clearance (CL) of acMMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Half-life (t1/2) of acMMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Volume of Distribution Under Steady-State Conditions (Vss) of acMMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Area Under the Plasma Concentration-Time Curve (AUC) for Unconjugated Monomethyl Auristatin E (MMAE) | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Maximum Observed Plasma Concentration (Cmax) for Unconjugated MMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Total Clearance (CL) of Unconjugated MMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Half-life (t1/2) of Unconjugated MMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Volume of Distribution Under Steady-State Conditions (Vss) of Unconjugated MMAE | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Monotherapy arm: Pre-infusion, 0.5, 4, hours after end of infusion on Cycle 1 Day 1; at Cycle 1 Days 2, 4 (or 5), 8, 11 (or 12), 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 2-4 Day 1, Cycle 2-4 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2 and 4 months after ET.
  Combination therapy arm: Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 2; at Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 2, Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, Cycle 12, and every 4th cycle thereafter up to ET visit.
  Pre-infusion = 0-4 hours before infusion; infusion duration = 90 minutes for first infusion and 30 minutes for other infusions, ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Obinutuzumab Serum Concentration | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 1; Cycle 1 Days 4 (or 5); Pre-infusion and 0.5 hours after end of infusion on Cycle 1 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 1; Pre-infusion and 0.5 hours after end of infusion on Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2, 4, 6 months after ET.
  Pre-infusion = 0-4 hours before infusion; infusion rate = 50 milligrams per hour initially (to be adjusted in case of reactions), ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Rituximab Serum Concentration | Pre-infusion on Cycle 1 Day 1 up to 1 year (detailed timeframe is provided in outcome description section)
  Pre-infusion, 0.5 hours after end of infusion on Cycle 1 Day 1; Cycle 1 Days 4 (or 5), 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycle 2 Day 1; Pre-infusion and 0.5 hours after end of infusion on Cycles 3-4 Day 1; Cycles 3-4 Days 8, 15; Pre-infusion and 0.5 hours after end of infusion on Cycles 5-8, 12, and every 4th cycle thereafter up to ET visit; 2, 4, 6 months after ET.
  Pre-infusion = 0-4 hours before infusion; infusion rate = 50 milligrams per hour initially (to be adjusted in case of reactions), ET = 30 days after last dose (up to 1 year), cycle length = 21 days.
Percentage of Participants with Anti-DCDS0780A Antibodies | Baseline up to 2 to 4 months after last dose (up to 16 months)
Absolute Lymphocyte Count | Cycle 1 Day 1 (Baseline); Day 1 of Cycles 4, 8, and every 4 cycles thereafter up to ET visit (up to 1 year); follow-up (up to 3.4 years)
Change from Baseline in Intra-Patient Absolute Lymphocyte Counts | Cycle 1 Day 1 (Baseline); Day 1 of Cycles 4, 8, and every 4 cycles thereafter up to ET visit (up to 1 year); follow-up (up to 3.4 years)
Time to CD19+ B-Cell Count Recovery to Baseline Value | Cycle 1 Day 1 (Baseline); Day 1 of Cycles 4, 8, and every 4 cycles thereafter up to ET visit (up to 1 year); follow-up (up to 3.4 years)
Percentage of Participants with Best Overall Response of Complete Response (CR) or Partial Response (PR) Assessed According to Lugano Classification | Baseline up to first occurrence of disease progression or death from any cause within 30 days after the last dose of study drug (up to 1 year)
Duration of Response Assessed According to Lugano Classification | From the first occurrence of a documented objective response (CR or PR) to the time of relapse or death from any cause (up to 1 year)
Progression-Free Survival (PFS) Assessed According to Lugano Classification | Baseline up to first occurrence of disease progression or death from any cause within 30 days after the last dose of study drug (up to 1 year)
Relative Dose Intensity (DI) Calculated as Ratio of Amount of Drug Actually Administered to the Amount Planned | Baseline up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Medical Center of Aurora; Rocky Mountain Cancer Centers, Aurora, Colorado
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Sarasota (North Catttlemen Rd), Sarasota, Florida
  - New York University Cancer Cen, New York, New York
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon